CLINICAL TRIAL: NCT02159508
Title: An Intervention Study Comparing Intensive Nutrition Counselling With On-demand Counselling in Patients With Head and Neck Cancer Undergoing Chemoradiotherapy
Brief Title: Intensive Nutrition Counselling in Patients With Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Helena Orell-Kotikangas, Dietitian, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 322-E9-05
Record Dates: First submitted 2014-04-29; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-05

CONDITIONS: Head and Neck Squamous Cell Cancer
Keywords: nutritional status; nutritional intervention; handgrip strength; patient-generated subjective global assessment; chemoradiotherapy; survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualised on-demand counselling (No Intervention): Individualized on-demand counselling group was assigned to receive baseline nutritional counselling, that consisted of one dietetic consultation before (chemo)radiotherapy. During (chemo)radiotherapy on-demand counselling group patients received further counselling only on demand.
- Intensive nutritional counselling (Experimental): Intensive nutritional counselling consisted of protocolled counselling given by a dietitian once at baseline and on the 2nd and 4th week of treatment and at the end of chemoradiotherapy.
  Interventions: Behavioral: Nutritional counselling

INTERVENTIONS:
Behavioral: Nutritional counselling — In both study arms, daily estimated energy requirements were calculated from the basal energy requirements according to WHO multiplied by a 1.5 activity factor and protein requirement (g/day) was calculated multiplying ideal body weight (defined as BMI 22) by 1.2 to 1.5.
  Arms: Intensive nutritional counselling

SUMMARY:
The purpose of this study is to assess the effect of a pre-planned patient-adjusted intensive nutritional counselling given by a dietitian several times during (chemo)radiotherapy vs. individualized nutritional counselling given by a dietitian once in the beginning of (chemo)radiotherapy and thereafter on-demand in patients with head and neck squamous cell cancer.

DETAILED DESCRIPTION:
* A sample size of 102 patients was identified to achieve 30% reduction in prevalence of malnutrition at the end of treatment (50% to 20%), with a significance value of 5% (p < 0.05), 90% power. The second calculation was for a sample size of 88 patients for 30% reduction in prevalence of malnutrition at the end of treatment (50% to 20%) with the significance value 5% (p<0.05), 85% power and effect size 70%. Based on these numbers, our aim is to recruit 100 patients, with the assumption that 12% patients would be lost to follow up.
* Randomization will be performed by the minimization procedure with the Minim Program® (http://www-users.york.ac.uk/~mb55/guide/randsery.htm). The allocation will be done according to the following criteria: 1) Stage I-II vs. Stage III-IV; 2) age <65 vs. >=65 year; 3) Body Mass Index <20 vs. >=20 kg/m2 and 4) tumour location (oral cavity-oropharynx-tonsils vs. hypopharynx-larynx vs. nasopharynx).
* Adverse events of chemoradiotherapy will be classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events-3.0 (CTCAE v3.0)
* Nutritional status will be assessed by patient-generated subjective global assessment, nutritional risk screening-2002, upper-arm anthropometry (MAC, triceps skinfold thickness, MAMA), Bio-impedance, hand grip strength and weight loss.
* Survival: overall survival, disease-specific survival and disease-free survival are calculated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary locally advanced squamous cell carcinoma of the oral cavity, pharynx, nasopharynx or larynx

Exclusion Criteria:

* renal function impairment
* liver insufficiency
* heart failure
* pulmonal impairment
* Chronic obstructive pulmonary disease
* cognitive impairment
* previous cancer in any location
* terminal stage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | 6 months
  Nutritional status was assessed by patient-generated subjective global assessment and anthropometry.

SECONDARY OUTCOMES:
Survival | 5 year
  Overall survival (OS) is defined as the time interval between the date of the randomization (i.e. at diagnosis) and the date of the last visit or death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Mäkitie, Professor, Study Director — Helsinki University Central Hospital
Locations (1):
- Department of Otolaryngology - Head & Neck Surgery, Helsinki University Central Hospital and University of Helsinki, Helsinki, HUS, Finland

REFERENCES:
- [Background] Isenring EA, Bauer JD, Capra S. Nutrition support using the American Dietetic Association medical nutrition therapy protocol for radiation oncology patients improves dietary intake compared with standard practice. J Am Diet Assoc. 2007 Mar;107(3):404-12. doi: 10.1016/j.jada.2006.12.007. PMID 17324657
- [Background] Ottery FD. Definition of standardized nutritional assessment and interventional pathways in oncology. Nutrition. 1996 Jan;12(1 Suppl):S15-9. doi: 10.1016/0899-9007(96)90011-8. PMID 8850213
- [Background] White JV, Guenter P, Jensen G, Malone A, Schofield M; Academy of Nutrition and Dietetics Malnutrition Work Group; A.S.P.E.N. Malnutrition Task Force; A.S.P.E.N. Board of Directors. Consensus statement of the Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition: characteristics recommended for the identification and documentation of adult malnutrition (undernutrition). J Acad Nutr Diet. 2012 May;112(5):730-8. doi: 10.1016/j.jand.2012.03.012. Epub 2012 Apr 25. PMID 22709779
- [Derived] Orell H, Schwab U, Saarilahti K, Osterlund P, Ravasco P, Makitie A. Nutritional Counseling for Head and Neck Cancer Patients Undergoing (Chemo) Radiotherapy-A Prospective Randomized Trial. Front Nutr. 2019 Mar 18;6:22. doi: 10.3389/fnut.2019.00022. eCollection 2019. PMID 30937304